CLINICAL TRIAL: NCT04305873
Title: Effect of Exercise-induced Hypoxemia on Cytokine and Stress Hormone Responses Among Endurance-trained Athletes
Brief Title: Cytokine and Stress Hormone Responses to Exercise-induced Hypoxemia Among Endurance-trained
Status: Enrolling by invitation | Type: Observational
Sponsor: Gepner Yftach (Other)
Responsible Party: Sponsor-Investigator, Gepner Yftach, Principal Investigator,, Tel Aviv University
Organization: Tel Aviv University (Other)
Other Study IDs: EIAH1
Record Dates: First submitted 2020-03-04; First posted 2020-03-12 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Exercise-induced Arterial Hypoxemia
Keywords: High intensity exercise; Endurance; Athletes; Desaturation; Stress response; Inflammatory markers
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EIAH athletes: Athletes with arterial oxyhemoglobin saturation at maximal exercise during a graded exercise test <93%
- Non-EIAH athletes: Athletes with arterial oxyhemoglobin saturation at maximal exercise during a graded exercise test >95%
- Intermediate EIAH athletes: Athletes with arterial oxyhemoglobin saturation at maximal exercise during a graded exercise test of 93-95%

SUMMARY:
It is well documented that exercise-induced arterial hypoxemia (EIAH) is highly prevalent among endurance-trained athletes performing heavy intensity exercise, regardless of sex and age. Although it has been shown that a drop in arterial oxyhemoglobin saturation (SaO2) during exercise (i.e. EIAH) negatively affects aerobic capacity measures such as VO2max and time trial performance, there remains a gap in the literature as to the physiological consequences of EIAH, and specifically acute cytokines and stress-related responses to hypoxemia during exercise. Exposure to hypoxic environments in which SaO2 is reduced and exercise can each, independently, alter/activate various pro- and anti-inflammatory markers and increases stress hormones. It follows then that EIAH athletes could be more susceptible to, and encounter more frequently, episodes of elevated levels of inflammatory cytokines and an exaggerated stress response than non-EIAH athletes; however, to the best of the investigators knowledge, this is yet to be confirmed. Therefore, it is hypothesized that highly trained endurance athletes who develop EIAH will experience more pronounced increases in inflammatory cytokines and stress hormones following a bout of heavy intensity exercise compared to athletes without EIAH.

DETAILED DESCRIPTION:
Fifty highly trained endurance runners (men and women, age: 18-35 years) will be recruited for this study. The first testing session will serve as a screening tool to determine subject eligibility. Following the first testing sessions subjects will be divided into EIAH or non-EIAH groups based on SaO2 at VO2max (EIAH < 93%, non-EIAH > 95%; Dempsey and Wagner criteria). Subjects with intermediate SaO2 (93-95% at VO2max) values will be included in the study for correlational analyses only.

All subjects will be advised orally, and in writing, as to the nature of the experiments and will give written, informed consent to the study protocol.

Study Design & protocol:

Subjects will be asked to visit the Exercise Performance Laboratory at the Sylvan Adams Sports Institute on three occasions. During the first visit subject will perform resting pulmonary function tests (PFTs) followed by a graded exercise test to exhaustion on either a motorized-treadmill for the determination of VO2max, degree of EIAH (SaO2 at VO2max) and maximal heart rate (HRmax). On the second visit, subjects will perform PFTs, followed by a brief warm-up run for 10 min at a moderate intensity equivalent to 60% of HRmax, as obtained from the incremental test and a 30-min trial at either half-marathon pace (HM30), designed to simulate a tempo workout often practiced by endurance runners. The third visit, conducted 24 hours after the 30-min trial, will include a blood draw only.

ELIGIBILITY:
Inclusion Criteria:

* 1) Physically active (minimum of 50 km running/week) and maximal oxygen consumption > 55 and 50 ml/kg-1/min-1 for men and women, respectively.
* 2) classified as low risk based on a medical questionnaire, body mass index and non-smoking status.
* 3) No history of pulmonary, metabolic and/or cardiovascular disease.
* 4) normal pulmonary function as defined by a ≥ 80% of predicted forced vital capacity (FVC), forced expired volume in one second (FEV1) and FEV1/FVC according the American Thoracic Society standards.

Exclusion Criteria:

* Smoking and/or any pulmonary, metabolic and/or cardiovascular disease.
* maximal oxygen consumption lower than set criteria.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Highly endurance trained athletes who have run a half marathon or marathon in the past.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cytokines | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
  Changes in Inflammatory cytokines (e.g. IL-6, IL-1b, IL-ra, IL-10)
Inflammatory cytokine | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
  Changes in Inflammatory cytokine TNF-a
Changes in Cortisol level | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
  Stress hormones
Changes in epinephrine level | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
  Stress hormones
Changes in norepinephrine level | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
  Stress hormones

SECONDARY OUTCOMES:
Changes in number of Neutrophiles | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
Changes in number of lymphocytes | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
Changes in number of monocytes | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
Immune markers | Changes from baseline to immediately, 2 hour and 24 hour post 30 minutes run at half marathon pace (HM30)
  Changes in basophiles count (number of)

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

REFERENCES:
- [Background] Babb TG. Exercise ventilatory limitation: the role of expiratory flow limitation. Exerc Sport Sci Rev. 2013 Jan;41(1):11-8. doi: 10.1097/JES.0b013e318267c0d2. PMID 23038244
- [Background] Bayliss DA, Millhorn DE. Central neural mechanisms of progesterone action: application to the respiratory system. J Appl Physiol (1985). 1992 Aug;73(2):393-404. doi: 10.1152/jappl.1992.73.2.393. PMID 1399957
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Behan M, Kinkead R. Neuronal control of breathing: sex and stress hormones. Compr Physiol. 2011 Oct;1(4):2101-39. doi: 10.1002/cphy.c100027. PMID 23733699
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Chapman RF, Emery M, Stager JM. Extent of expiratory flow limitation influences the increase in maximal exercise ventilation in hypoxia. Respir Physiol. 1998 Jul;113(1):65-74. doi: 10.1016/s0034-5687(98)00043-7. PMID 9776552
- [Background] Duke JW, Stickford JL, Weavil JC, Chapman RF, Stager JM, Mickleborough TD. Operating lung volumes are affected by exercise mode but not trunk and hip angle during maximal exercise. Eur J Appl Physiol. 2014 Nov;114(11):2387-97. doi: 10.1007/s00421-014-2956-0. Epub 2014 Aug 2. PMID 25085604
- [Background] Pearman T, Yanez B, Peipert J, Wortman K, Beaumont J, Cella D. Ambulatory cancer and US general population reference values and cutoff scores for the functional assessment of cancer therapy. Cancer. 2014 Sep 15;120(18):2902-9. doi: 10.1002/cncr.28758. Epub 2014 May 22. PMID 24853866
- [Background] Johnson BD, Saupe KW, Dempsey JA. Mechanical constraints on exercise hyperpnea in endurance athletes. J Appl Physiol (1985). 1992 Sep;73(3):874-86. doi: 10.1152/jappl.1992.73.3.874. PMID 1400051
- [Background] Johnson BD, Weisman IM, Zeballos RJ, Beck KC. Emerging concepts in the evaluation of ventilatory limitation during exercise: the exercise tidal flow-volume loop. Chest. 1999 Aug;116(2):488-503. doi: 10.1378/chest.116.2.488. PMID 10453881
- [Background] McClaran SR, Harms CA, Pegelow DF, Dempsey JA. Smaller lungs in women affect exercise hyperpnea. J Appl Physiol (1985). 1998 Jun;84(6):1872-81. doi: 10.1152/jappl.1998.84.6.1872. PMID 9609779
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Weavil JC, Duke JW, Stickford JL, Stager JM, Chapman RF, Mickleborough TD. Endurance exercise performance in acute hypoxia is influenced by expiratory flow limitation. Eur J Appl Physiol. 2015 Aug;115(8):1653-63. doi: 10.1007/s00421-015-3145-5. Epub 2015 Mar 13. PMID 25761731
- [Background] Romer LM, Dempsey JA, Lovering A, Eldridge M. Exercise-induced arterial hypoxemia: consequences for locomotor muscle fatigue. Adv Exp Med Biol. 2006;588:47-55. doi: 10.1007/978-0-387-34817-9_5. PMID 17089878
- [Background] Amann M, Eldridge MW, Lovering AT, Stickland MK, Pegelow DF, Dempsey JA. Arterial oxygenation influences central motor output and exercise performance via effects on peripheral locomotor muscle fatigue in humans. J Physiol. 2006 Sep 15;575(Pt 3):937-52. doi: 10.1113/jphysiol.2006.113936. Epub 2006 Jun 22. PMID 16793898
- [Background] Dempsey JA, Wagner PD. Exercise-induced arterial hypoxemia. J Appl Physiol (1985). 1999 Dec;87(6):1997-2006. doi: 10.1152/jappl.1999.87.6.1997. PMID 10601141
- [Background] Constantini K, Tanner DA, Gavin TP, Harms CA, Stager JM, Chapman RF. Prevalence of Exercise-Induced Arterial Hypoxemia in Distance Runners at Sea Level. Med Sci Sports Exerc. 2017 May;49(5):948-954. doi: 10.1249/MSS.0000000000001193. PMID 28009787
- [Background] Dominelli PB, Molgat-Seon Y, Griesdale DEG, Peters CM, Blouin JS, Sekhon M, Dominelli GS, Henderson WR, Foster GE, Romer LM, Koehle MS, Sheel AW. Exercise-induced quadriceps muscle fatigue in men and women: effects of arterial oxygen content and respiratory muscle work. J Physiol. 2017 Aug 1;595(15):5227-5244. doi: 10.1113/JP274068. Epub 2017 Jun 19. PMID 28524229
- [Background] Richards JC, McKenzie DC, Warburton DE, Road JD, Sheel AW. Prevalence of exercise-induced arterial hypoxemia in healthy women. Med Sci Sports Exerc. 2004 Sep;36(9):1514-21. doi: 10.1249/01.mss.0000139898.30804.60. PMID 15354032
- [Background] Hopkins SR, Barker RC, Brutsaert TD, Gavin TP, Entin P, Olfert IM, Veisel S, Wagner PD. Pulmonary gas exchange during exercise in women: effects of exercise type and work increment. J Appl Physiol (1985). 2000 Aug;89(2):721-30. doi: 10.1152/jappl.2000.89.2.721. PMID 10926659
- [Background] Hopkins SR. Exercise induced arterial hypoxemia: the role of ventilation-perfusion inequality and pulmonary diffusion limitation. Adv Exp Med Biol. 2006;588:17-30. doi: 10.1007/978-0-387-34817-9_3. PMID 17089876
- [Background] Rice AJ, Thornton AT, Gore CJ, Scroop GC, Greville HW, Wagner H, Wagner PD, Hopkins SR. Pulmonary gas exchange during exercise in highly trained cyclists with arterial hypoxemia. J Appl Physiol (1985). 1999 Nov;87(5):1802-12. doi: 10.1152/jappl.1999.87.5.1802. PMID 10562625